CLINICAL TRIAL: NCT00412880
Title: An Open-label Phase II Trial to Investigate the Efficacy, Safety, and Pharmacokinetics of a Single Dose of 200 mg i.v. BI 2536 Administered Every 21 Days in Patients With Sensitive Relapse Small Cell Lung Cancer
Brief Title: BI 2536 Second Line Monotherapy in SCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1216.11
Record Dates: First submitted 2006-12-18; First posted 2006-12-19 (Estimated); Results first posted 2022-05-31 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-05

CONDITIONS: Carcinoma, Small Cell
MeSH Terms: conditions — Carcinoma, Small Cell | interventions — BI 2536

ARMS (1):
- BI 2536 (Experimental): Total Patients
  Interventions: Drug: BI 2536

INTERVENTIONS:
Drug: BI 2536 — Intravenous Infusion

SUMMARY:
Open label, uncontrolled Phase II trial to assess the efficacy and safety of BI 2536 in second line treatment in sensitive-relapse SCLC patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed, -sensitive-relapse- SCLC defined by a relapse 60 days or more after cessation of prior first-line chemotherapy.
* Patients with at least one measurable lesion, with longest diameter to be recorded as 20 mm or greater.
* Life expectancy of at least three months and ECOG performance score of 2 or less and written informed consent that must be consistent with ICH-GCP Guidelines.

Exclusion Criteria:

* More than one prior regimen of chemotherapy, mixed small cell/large cell or combined small cell histology.
* Symptomatic brain metastases or leptomeningeal disease
* Patients with ascites, patients who have any other life-threatening illness or organ system dysfunction, or other malignancies diagnosed within the past five (5) years (other than non melanomatous skin cancer)
* Absolute neutrophil count (ANC) <1,500/µl, platelet count <100,000/µl, or hemoglobin <9 mg/dl
* Total bilirubin >1.5 x ULN, aspartame amino transferase (AST) and/or alanine amino transferase (ALT) >2.5 x ULN, or aspartate amino transferase (AST) and/or alanine amino transferase (ALT) >5 x ULN in case of known liver metastases, serum creatinine >2.0 mg/dl (>176 µmol/L, SI Unit equivalent)
* Chemo-, hormone- (other than Megace®) or immunotherapy within the past 4 weeks or within less than 4 half-life times of the previous drug prior to treatment with the trial drug
* Radiation therapy within the past 2 weeks prior to or during treatment with the trial drug
* Patients with any serious active infection (i.e., requiring an IV antibiotic, antifungal, or antiviral agents), patients with known HIV, hepatitis-B or -C infection
* Known or suspected active drug or alcohol abuse
* Treatment with any other investigational drug within the past 4 weeks or within less than 4 half-life times of the investigational drug
* Patients with a known pre-existing coagulopathy or requiring therapeutic anticoagulation with warfarin (Coumadin ®)
* Patients with neuropathy (sensory or motor) CTCAE 3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-02-14 (Actual); Primary Completion 2008-06-30 (Actual); Study Completion 2008-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (10):
- United States (9):
  - 1216.11.007 Boehringer Ingelheim Investigational Site, Fayetteville, Arkansas
  - 1216.11.003 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 1216.11.006 Boehringer Ingelheim Investigational Site, Evanston, Illinois
  - 1216.11.002 Boehringer Ingelheim Investigational Site, Boston, Massachusetts
  - 1216.11.005 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 1216.11.001 Boehringer Ingelheim Investigational Site, Chapel Hill, North Carolina
  - 1216.11.011 Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - 1216.11.010 Boehringer Ingelheim Investigational Site, Greenville, South Carolina
  - 1216.11.012 Boehringer Ingelheim Investigational Site, Seattle, Washington
- 1216.11.009 Alberta Cancer Board, Edmonton, Alberta, Canada

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is an open-label Phase II trial to investigate the efficacy, safety, and pharmacokinetics of a single dose of 200 mg i.v. BI 2536 administered every 21 days in patients with sensitive relapse small cell lung cancer using an uncontrolled, Gehan two-stage trial design with an early stopping rule based on patient response.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- BI 2536 200 mg: Patients received a single intravenous infusion of 200 milligram (mg) BI 2536 on day 1 of each 21 day treatment cycle. Beyond the second treatment cycle patients may either be treated with the original dose or may receive a higher dose in case of clinical benefit and good tolerability. BI 2536 dosing can be increased in steps of 50 mg. Dose escalations may be repeated after every other course.
Period: Overall Study
Arm/Group | BI 2536 200 mg
Started | 23
Completed | 0
Not Completed | 23
Not completed — Withdrew, overdose of study treatment | 1
Not completed — Consent withdrawn | 1
Not completed — Adverse Event | 1
Not completed — Progressive disease | 20

BASELINE CHARACTERISTICS:
Population: Treated set (TS): includes all patients who were documented to have taken at least one application of BI 2536.
Arm/Group | BI 2536 200 mg
Number analyzed (Participants) | 23
Age, Continuous [Median (Full Range); unit: years] | 60.0 [35 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Tumor Response
Description: Objective tumor response by investigator was assessed for patients who completed at least two courses of BI 2536 treatment. Tumor images from CT (computed tomography) scan and MRI (magnetic resonance imaging) were evaluated using Response evaluation criteria in solid tumors (RECIST) criteria to determine best tumor response. Objective response (OR) was defined as either: complete response (CR, disappearance of all target lesions) or partial response (PR, at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter).
Time Frame: Scans during screening (day -28 till day 0) and day 1 of every other (even numbered) 21 day treatment cycle. Up to 40 weeks.
Population: Treated set (TS): includes all patients who were documented to have taken at least one application of BI 2536. Four patients were excluded from this endpoint due to not having completed two treatment cycles (21 days each).
Measure: Count of Participants; unit: Participants
Arm/Group | BI 2536 200 mg
Number analyzed (Participants) | 19
Participants
  Complete response | 0
  Partial response | 0

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression free survival (PFS) was defined as the duration of time from start of treatment to time of progression (or death any cause). Patients who did not experience progression or death during the trial were censored at the date of last tumor assessment visit at which the patient was evaluated and did not experience progressive disease. Patients who dropped out before any evaluation of response, radiological, clinical, or pathological, were censored at the start of treatment. Progressive Disease (PD) was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: as for outcome 1
Population: Treated set (TS): includes all patients who were documented to have taken at least one application of BI 2536.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | BI 2536 200 mg
Number analyzed (Participants) | 23
days | 43 [40 to 50]

3. Secondary Outcome: Overall Survival
Description: Overall survival (OS) was reported as number of participants with event. Overall survival is the time from first treatment to death. In case there was no occurrence of death or progression during follow-up, the time was censored.
  Median survival time was not calculated due to the low number of deaths in the trial.
Time Frame: From the start of treatment till death or discontinuation, up to 36 weeks.
Population: Treated set (TS): includes all patients who were documented to have taken at least one application of BI 2536..
Measure: Count of Participants; unit: Participants
Arm/Group | BI 2536 200 mg
Number analyzed (Participants) | 23
Participants | 5

4. Secondary Outcome: Duration of Overall Response
Description: The duration of overall objective response (OR) was measured from the time measurement criteria were met for complete response (CR) or partial response (PR) (whichever was first recorded) until the first date that recurrent or progressive disease was objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started) or death any cause. OR is defined as either: CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter).
Time Frame: as for outcome 1
Population: Analysis of duration of overall response was not conducted, as there were no responders
Arm/Group | BI 2536 200 mg
Number analyzed (Participants) | 0

5. Secondary Outcome: Occurrence and Intensity of Adverse Events Graded According to CTCAE
Description: Occurrence and intensity of adverse events graded according to common terminology criteria of adverse event (CTCAE) version 3.0.
Time Frame: From the start of treatment till the last infusion + 21 days, up to 36 weeks.
Population: Treated set (TS): includes all patients who were documented to have taken at least one application of BI 2536.
Measure: Count of Participants; unit: Participants
Arm/Group | BI 2536 200 mg
Number analyzed (Participants) | 23
Participants
  CTCAE grade 1 | 1
  CTCAE grade 2 | 4
  CTCAE grade 3 | 8
  CTCAE grade 4 | 6
  CTCAE grade 5 | 2

6. Secondary Outcome: Number of Participants With Dose Limiting Toxicity
Description: Number of Participants with Dose Limiting Toxicity. Dose limiting toxicity was defined as:
  * drug related CTCAE Grade 3 or greater non-hematological toxicity (excluding untreated nausea, vomiting or diarrhea)
  * drug related CTCAE Grade 4 neutropenia for 7 or more days or complicated by infection
  * CTCAE Grade 4 thrombocytopenia.
Time Frame: From the start of treatment till the last treatment + 21 days, up to 36 weeks.
Population: Treated set (TS): includes all patients who were documented to have taken at least one application of BI 2536.
Measure: Count of Participants; unit: Participants
Arm/Group | BI 2536 200 mg
Number analyzed (Participants) | 23
Participants | 4

7. Secondary Outcome: Number of Participants With an Increase in CTC Grade Classification for Hematological and Clinical Chemistry Laboratory Measures
Description: Number of participants with an increase in common terminology criteria (CTC) Grade classification for hematological and clinical chemistry laboratory measures. Changes from Baseline in laboratory measures were classified according to CTC Grades 1-4. Results summarizes the number of patients who had a change in laboratory value that represented an increase in CTC Grade classification during the study (based on maximum Grade).
Time Frame: From the start of treatment till the last treatment + 21 days, up to 36 weeks.
Population: Treated set (TS): includes all patients who were documented to have taken at least one application of BI 2536.
Measure: Count of Participants; unit: Participants
Arm/Group | BI 2536 200 mg
Number analyzed (Participants) | 23
Participants
  Lymphocytes: CTC Grade 1 | 3
  Lymphocytes: CTC Grade 2 | 4
  Lymphocytes: CTC Grade 3 | 6
  Lymphocytes: CTC Grade 4 | 1
  Lymphocytes: no increase in CTC grade | 9
  Neutrophil: CTC Grade 1 | 0
  Neutrophil: CTC Grade 2 | 4
  Neutrophil: CTC Grade 3 | 6
  Neutrophil: CTC Grade 4 | 11
  Neutrophil: no increase in CTC grade | 2
  Aspartate aminotransferase: CTC Grade 1 | 4
  Aspartate aminotransferase: CTC Grade 2 | 0
  Aspartate aminotransferase: CTC Grade 3 | 2
  Aspartate aminotransferase: CTC Grade 4 | 0
  Aspartate aminotransferase: no increase in CTC grade | 17
  Alanine aminotransferase: CTC Grade 1 | 4
  Alanine aminotransferase: CTC Grade 2 | 1
  Alanine aminotransferase: CTC Grade 3 | 1
  Alanine aminotransferase: CTC Grade 4 | 0
  Alanine aminotransferase: no increase in CTC grade | 17
  Haemoglobin: CTC Grade 1 | 5
  Haemoglobin: CTC Grade 2 | 9
  Haemoglobin: CTC Grade 3 | 1
  Haemoglobin: CTC Grade 4 | 1
  Haemoglobin: no increase in CTC grade | 7
  Platelets: CTC Grade 1 | 10
  Platelets: CTC Grade 2 | 1
  Platelets: CTC Grade 3 | 3
  Platelets: CTC Grade 4 | 1
  Platelets: no increase in CTC grade | 8
  White blood cell count: CTC Grade 1 | 1
  White blood cell count: CTC Grade 2 | 8
  White blood cell count: CTC Grade 3 | 11
  White blood cell count: CTC Grade 4 | 3
  White blood cell count: no increase in CTC grade | 0
  Creatinine: CTC Grade 1 | 1
  Creatinine: CTC Grade 2 | 0
  Creatinine: CTC Grade 3 | 0
  Creatinine: CTC Grade 4 | 0
  Creatinine: no increase in CTC grade | 22
  Bilirubin, total: CTC Grade 1 | 0
  Bilirubin, total: CTC Grade 2 | 0
  Bilirubin, total: CTC Grade 3 | 2
  Bilirubin, total: CTC Grade 4 | 0
  Bilirubin, total: no increase in CTC grade | 21

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the start of treatment till the last treatment + 21 days, up to 36 weeks. All-Cause Mortality was collected from the start of treatment till death or discontinuation, up to 36 weeks.
Description: Treated set (TS): includes all patients who were documented to have taken at least one application of BI 2536.
Arm/Group | BI 2536 200 mg
All-Cause Mortality (participants affected / at risk) | 5/23
Serious Adverse Events (participants affected / at risk) | 5/23
Other Adverse Events (participants affected / at risk) | 21/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BI 2536 200 mg (N=23)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Disease progression (General disorders) | 1
Sepsis (Infections and infestations) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 2536 200 mg (N=23)
Anaemia (Blood and lymphatic system disorders) | 6
Leukopenia (Blood and lymphatic system disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 5
Constipation (Gastrointestinal disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 7
Stomatitis (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 6
Fatigue (General disorders) | 9
Pain (General disorders) | 3
Pyrexia (General disorders) | 2
Upper respiratory tract infection (Infections and infestations) | 2
White blood cell count decreased (Investigations) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4
Dizziness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 2
Hallucination (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 2
Hypotension (Vascular disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 2

LIMITATIONS AND CAVEATS:
The criteria for expanding the trial to the second stage were not achieved and the trial was stopped early per trial design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.